CLINICAL TRIAL: NCT04737707
Title: Dialectical Behavior Therapy for Adults With Autism Spectrum Disorders Without Intellectual Disability: a Randomized Controlled Trial
Brief Title: Dialectical Behavior Therapy for Adults With Autism Spectrum Disorders
Acronym: Autisemo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8108
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behavior Therapy (DBT) (Experimental): Psychotherapy (duration 5 months) will begin within a maximum of 1 month (the time to set up the group) and will be accompanied by individual follow-up. Evaluations will be carried out within 6 months of the end of the psychotherapy in order to measure its effects.
  Interventions: Other: Dialectical Behavior Therapy (DBT)
- Therapy (Other): waiting list for 5 months before starting psychotherapy (duration 5 months). During this time, the patient can continue your usual therapeutic follow-ups. Likewise, assessments will be carried out within 6 months after the end of the psychotherapy in order to measure its effects. the patient will thus benefit from DBT regardless of the group.
  Interventions: Other: Dialectical Behavior Therapy (DBT)

INTERVENTIONS:
Other: Dialectical Behavior Therapy (DBT) — Dialectical Behavior Therapy (DBT)

SUMMARY:
Dialectical Behavior Therapy (DBT; Linehan, 1993) effectively diminishes emotion dysregulation and self-harm behaviors in a number of disorders. However, to our knowledge, no studies have investigated the efficacy of DBT to treat emotional dysregulation associated with self-harm and suicidal behaviors in adults with ASD without intellectual disability. This randomized controlled study trial aims to assess the efficacy of a 5-month DBT intervention in adults with ASD without intellectual disability who present with self-harm and/or suicidal behaviors.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* ASD diagnosis according to the DSM-5
* IQ ≥ 70
* Suicidal ideas, suicidal attempts and/or self-harm behaviors 6 months prior to the inclusion
* Able to understand and consent to the research aims
* Membership in a health insurance fund

Exclusion Criteria:

* complete hospitalization
* ongoing CBT or DBT
* past DBT
* schizophrenia disorders
* under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | baseline
  The minimum value of the DERS scale is 0 and the maximum is 180. The higher the scores, the more severe the deregulation.
Difficulties in Emotion Regulation Scale (DERS) | at the end of therapy (5 months)
  The minimum value of the DERS scale is 0 and the maximum is 180. The higher the scores, the more severe the deregulation.
Difficulties in Emotion Regulation Scale (DERS) | 11 months follow-up
  The minimum value of the DERS scale is 0 and the maximum is 180. The higher the scores, the more severe the deregulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de psychiatrie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiner L, Costache ME, Bemmouna D, Rabot J, Weibel S, Dubreucq M, Dubreucq J, Coutelle R. Emotion dysregulation is heightened in autistic females: A comparison with autistic males and borderline personality disorder. Womens Health (Lond). 2023 Jan-Dec;19:17455057231174763. doi: 10.1177/17455057231174763. PMID 37218688